CLINICAL TRIAL: NCT06727487
Title: OvS Breast: ENBI Project, Ovarian Suppression in Breast Cancer: Exercise, Nutrition and Behavioural Intervention Project
Brief Title: OvS Breast: Ovarian Suppression in Breast Cancer Interventions
Acronym: ENBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia Comillas (Other)
Collaborators: Hospital General Universitario Gregorio Marañon (Other); San Juan de Dios Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ENBI_2023
Record Dates: First submitted 2023-10-10; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Breast Neoplasms
Keywords: Physical Exercise; Nutritional advice; Psico-oncological support; Patient Report Outcomes
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1, control (Active Comparator): Group 1/Control: patients will receive the basic recommendations on healthy lifestyle habits indicated by the World Health Organization (WHO) through audiovisual material that they will receive via email. An explanatory video and a document with WHO guidelines will be included (https://apps.who.int/iris/bitstream/handle/10665/337004/9789240014817-spa.pdf).
  Interventions: Behavioral: Basic recommendations
- Group 2, experimental (Experimental): Group 2/ Exercise, nutrition, and psycho-oncological support: patients will carry out a cardiovascular and strength exercise program of moderate-high intensity at the facilities of the Exercise and Cancer Center organized in sessions of 60 to 75 minutes in duration, with a frequency of 2 days/week for 12 weeks; In addition, 3 sessions of nutritional counseling and 3 sessions of psycho-oncological intervention will be developed.
  Interventions: Behavioral: Physical exercise; Behavioral: Nutritional advice; Behavioral: Psycho-oncological support

INTERVENTIONS:
Behavioral: Basic recommendations — Daily basis activity counseling by WHO recommendations
  Arms: Group 1, control
Behavioral: Physical exercise — A complete program of active physical exercise of medium and high intensity
  Arms: Group 2, experimental
Behavioral: Nutritional advice — A complete program of nutritional counseling
  Arms: Group 2, experimental
Behavioral: Psycho-oncological support — A program related with a patient Psycho-oncological follow-up
  Arms: Group 2, experimental

SUMMARY:
The goal of this clinical trial is to compare a combined intervention based on physical exercise, nutritional control, and individualized psycho-oncological support can achieve weight control and maintain adequate body composition in premenopausal women with localized BC with ER and/or PR expression who receive aLHRH in combination with TAM or AI as part of adjuvant treatment.

The study's primary objectives are to evaluate the impact of the combined intervention on weight reduction and favorable modification of body composition in terms of reduction in body fat and increase in lean mass.

The secondary objectives aim to evaluate the impact of the combined intervention program on CRF, heart rate (HR), capillary lactate levels, upper and lower body strength, physical functionality, and patient-reported outcomes (PROs). (exercise level, asthenia, self-perception, anxiety and depression), blood count and biochemistry values that could be modified, nutritional situation, and side effects of treatments.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common and incident neoplasia in women in Spain and is the third cause of cancer death after lung and colorectal cancer. In turn, BC with hormone receptor expression is the most common and corresponds to approximately 75% of BC cases.

Suppression of ovarian function combined with endocrine treatment (gonadotropin-releasing hormone analog (LHRH) associated with tamoxifen (TAM) or aromatase inhibitors (AI)) has demonstrated a benefit in terms of relapse-free survival (PFS) and overall survival (OS) in premenopausal women diagnosed with localized BC with estrogen receptor (ER) and progesterone (PR) expression. This benefit is mainly focused on patients diagnosed at younger ages (under 45 years) and those with other clinical-pathological factors that imply an exceptionally high risk of relapse.

Despite their benefits, the adverse effects of these treatments are not trivial and include significant toxicities in the cardiorespiratory, metabolic, sexual, and emotional spheres. Metabolic alterations include unfavorable changes in body composition with increases in the percentage of fat and weight that can be observed already in the first months of treatment, which in turn is directly related to an increased risk of BC relapse in these patients.

Changes in body composition with increased fat and decreased muscle mass lead to a pro-inflammatory and dysfunctional state of the immune system, which in turn has been linked to the development of cardiovascular diseases and a worse oncological prognosis.

Scientific evidence suggests that nutritional interventions combined with physical exercise and adapted to physiological needs, the baseline physical level, and the adverse effects derived from the treatments can be safe and effective in achieving adequate weight control and body composition. All of this would favor restoring the immune system's functionality and increasing patients' cardiorespiratory capacity (CRF), which could ultimately translate into a better quality of life.

However, adherence to these programs is low for many reasons, and psycho-oncological support with behavioral interventions could favor adherence to them and stimulate changes in patients' lifestyles.

Despite the evidence, there is no scientific consensus regarding the dosage of exercise and the type of nutritional intervention that should be applied to patients with BC whose treatment includes suppression of ovarian function. In this sense, these interventions should be individualized and adapted to the characteristics of each patient, taking into account all the factors that could affect adherence to these programs.

This project has been designed as a pilot study to evaluate the impact of an intervention program incorporating physical exercise and nutritional control strategies adapted to the baseline situation and level of physical fitness of each premenopausal patient with localized BC on adjuvant treatment with ovarian function suppression.

HYPOTHESIS AND OBJECTIVES: combined intervention based on physical exercise, nutritional control, and individualized psycho-oncological support can achieve weight control and maintain adequate body composition in premenopausal women with localized BC with ER and PR expression who receive aLHRH in combination with TAM or AI as part of their adjuvant treatment.

The study's primary objectives are to evaluate the impact of the combined intervention on weight reduction and favorable modification of body composition in terms of reduction of body fat and increase of lean mass.

The secondary objectives aim to evaluate the impact of the combined intervention program on CRF, heart rate (HR), capillary lactate levels, upper and lower body strength, physical functionality, patient-reported outcomes (PROs) (exercise level, asthenia, self-perception, anxiety, and depression), blood count and biochemistry values that could be modified, nutritional status and side effects of the treatments.

The exploratory objectives, on the other hand, consist of evaluating the impact of the combined intervention on the levels of pro-inflammatory substances (C-reactive protein (CRP) and TNF-alpha) and anti-inflammatory substances (adiponectin) as well as on the levels of oncostatin M, a myokine whose release increases with exercise and seems to stimulate apoptosis and interfere with exercise.

ELIGIBILITY:
Inclusion Criteria:

* Women who have reached the age of majority and up to 45 years of age.
* Premenopausal status is defined clinically as a patient who maintains menstruation prior to the start of chemotherapy treatment if this has taken place.
* Confirmed histological diagnosis of infiltrating breast carcinoma with expression of ER and/or RP stage I to III.
* Loco-regional treatment with surgery and radiotherapy, if any, completed.
* Adjuvant treatment with drugs that suppress ovarian function (aLHRH) is ongoing and expected to be maintained for at least 4 months at the beginning of the study.
* Functional status according to the Eastern Cooperative Oncology Group (ECOG) scale 0-1.
* Ability to understand and agree to the Informed Consent in writing.

Exclusion Criteria:

* Presence of medical contraindications to perform physical exercise.
* Presence of any of the American Thoracic Society (ATS) criteria to perform a cardiovascular capacity test.
* Presence of active neoplastic disease: metastatic breast cancer or other active tumor diseases.
* Pregnancy or breastfeeding.
* Alcohol or other drug abuse (excluding smoking).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 30 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Combined intervention evaluation on weight control | 1 year
  A combined intervention based on physical exercise, nutritional control, and individualized psycho-oncological support can achieve weight control and maintain adequate body composition in premenopausal women with localized breast cancer expressing estrogen receptors and progesterone receptors who receive adjuvant treatment. The psycho-oncological intervention program aims to increase motivation to adhere to the physical exercise program and nutritional recommendations and maintain long-term healthy lifestyle habits.
Combined intervention evaluation in body composition | 1 year
  The variables weight, kilograms, fat mass, lean mass, and extracellular water will be obtained with the Tanita BC-601 Gold scale, including an impedance meter. The height, waist, and hip circumferences will be obtained with a tape measure. These measurements are necessary for calculating the BMI and the waist-high index (measure in centimeters). Weight and height will be combined to report BMI in kg/m^2 Units of measure: weight in kilograms, height in meters.

SECONDARY OUTCOMES:
Improve Quality of Life on Patient Report Outcomes | 1 year
  To evaluate the impact of the combined intervention program on patient-reported outcomes (PROs) (exercise level , asthenia, self-perception, anxiety and depression).
  The combination of several validated tests allows us to establish a balanced measure with the multi-professional approaches that care for the patient.
  Patient Reported Outcomes (PROs): These will be assessed and collected by completing validated questionnaires for this purpose.
  * Quality of life: EuroQoL-5D questionnaire
  * Fatigue: FACIT-Fatigue questionnaire
  * Level of physical activity: International Physical Activity Questionnaire (IPAQ)
  * Self-perception/self-esteem: Rosemberg Self-Esteem Scale
  * Anxiety and Depression: Hospital Anxiety and Depression Scale (HADS)
Nutritional Status follow-up | 1 year
  Nutritional status: It will be assessed using the following tools at the beginning, 6 weeks after the start of the intervention and at the end of the 12 weeks.The combination of several validated tests allows us to establish a balanced measure of the specific situation in each patient.
  * 3-day nutritional record
  * Predimed Mediterranean diet adherence questionnaire
  * WCRF/AICR recommendations compliance scale
Psycho-oncological assessment | 1 year
  Psycho-oncological assessment: It will be assessed with the following questionnaires that the patient will complete at the beginning and the end of the 12 weeks of intervention.
  The combination of several validated tests allows us to establish a measure that relates the emotional state with the variables of physical exercise The PANAS affectivity scale will have an additional intermediate evaluation six weeks after the start of the intervention.
  * PANAS affectivity scale
  * Transtheoretical model of change in physical exercise (CMTCEJ) questionnaire.
  * MOS social support questionnaire
Cardiorespiratory Fitness: Evaluation of physical activity performance | 1 year
  Evaluation of physical activity performance thought:
  -Cardiorespiratory fitness (CRF): The Bruce test will be evaluated to determine the maximum oxygen consumption (VO2max, milliliters/kilogram/minute). -Cardiac variability (HR at rest and maximum (beats/minute)): It will be measured with an HR receiver before the Bruce test (at rest) and at the time of finishing it (maximum effort)
Endurance performance: Evaluation of physical activity performance: | 1 year
  -Endurance performance (capillary lactate levels (millimoles/liter): They will be evaluated with a lactate analyzer at rest, at the time of finishing it (maximum effort), and two minutes after having finished it.
Strength: Evaluation of physical activity performance | 1 year
  -Strength: It will be evaluated using dynamometry of the upper and lower body, as well as with the squat test and shoulder press with load (kilograms mobilized and repetitions performed).
Physical functionality: Evaluation of physical activity performance | 1 year
  -Physical functionality: It will be measured with the maximum squat test in 30 seconds (number of repetitions) and 6-minute walk (maximum distance in meters that the patient can walk for 6 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Julio C de la Torre, Ph.D, Study Chair — Universidad Pontificia Comillas; Blanca Herrero López, MD, Principal Investigator — Hospital Universitario Gregorio Marañón; Soraya Casla Barrio, Ph.D, Study Director — Comillas Pontifical University
Locations (2):
- Spain (2):
  - Universidad Pontificia Comillas, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid

IPD SHARING:
Plan to Share IPD: Yes
A complete publication plan will be taken into account, covering everything from the protocol to the dissemination of the results in scientific journals and scientific forums, such as specialized conferences.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: Public access

REFERENCES:
- [Result] Francis PA, Pagani O, Fleming GF, Walley BA, Colleoni M, Lang I, Gomez HL, Tondini C, Ciruelos E, Burstein HJ, Bonnefoi HR, Bellet M, Martino S, Geyer CE Jr, Goetz MP, Stearns V, Pinotti G, Puglisi F, Spazzapan S, Climent MA, Pavesi L, Ruhstaller T, Davidson NE, Coleman R, Debled M, Buchholz S, Ingle JN, Winer EP, Maibach R, Rabaglio-Poretti M, Ruepp B, Di Leo A, Coates AS, Gelber RD, Goldhirsch A, Regan MM; SOFT and TEXT Investigators and the International Breast Cancer Study Group. Tailoring Adjuvant Endocrine Therapy for Premenopausal Breast Cancer. N Engl J Med. 2018 Jul 12;379(2):122-137. doi: 10.1056/NEJMoa1803164. Epub 2018 Jun 4. PMID 29863451
- [Result] Francis PA, Fleming GF, Lang I, Ciruelos EM, Bonnefoi HR, Bellet M, Bernardo A, Climent MA, Martino S, Bermejo B, Burstein HJ, Davidson NE, Geyer CE Jr, Walley BA, Ingle JN, Coleman RE, Muller B, Le Du F, Loibl S, Winer EP, Ruepp B, Loi S, Colleoni M, Coates AS, Gelber RD, Goldhirsch A, Regan MM; SOFT Investigators and the International Breast Cancer Study Group (a division of ETOP IBCSG Partners Foundation). Adjuvant Endocrine Therapy in Premenopausal Breast Cancer: 12-Year Results From SOFT. J Clin Oncol. 2023 Mar 1;41(7):1370-1375. doi: 10.1200/JCO.22.01065. Epub 2022 Dec 9. PMID 36493334
- [Result] Lu YS, Wong A, Kim HJ. Ovarian Function Suppression With Luteinizing Hormone-Releasing Hormone Agonists for the Treatment of Hormone Receptor-Positive Early Breast Cancer in Premenopausal Women. Front Oncol. 2021 Sep 14;11:700722. doi: 10.3389/fonc.2021.700722. eCollection 2021. PMID 34595110
- [Derived] Herrero Lopez B, Castellanos Montealegre M, Soulas C, Rufrancos BA, Garcia-Ontiveros Cuellar ML, Del Monte Millan M, Villarejo Lopez L, Lopez-Tarruella Cobo S, Jerez Gilarranz Y, Echavarria Diaz-Guardamino I, Jara P, Jimenez MM, Sanchez TM, Martinez Beltran MJ, de la Torre Montero JC, Casla Barrio S. Randomized pilot study of an individualized multimodal exercise, nutrition, and behavior intervention in breast cancer patients treated with ovarian function suppression: protocol proposal for The OvS Breast ENBI Project. Front Oncol. 2025 Oct 27;15:1622622. doi: 10.3389/fonc.2025.1622622. eCollection 2025. PMID 41220947
- See also: Cancer epidemiology in Spain — https://seom.org/images/Las_cifras_del_Cancer_en_Espana_2023.pdf